CLINICAL TRIAL: NCT02882230
Title: Prospective Evaluation of Neurologic and Psychiatric Adverse Events of Rilpivirine, Elvitegravir, or Dolutegravir in a Real Life Setting
Brief Title: Evaluation of Neurologic and Psychiatric Adverse Events of Several Antiretroviral Drugs in Real Life Setting
Acronym: NEPAL
Status: Terminated | Type: Observational
Why Stopped: Unfavourable opinion of ethical comittee for Amendment Nr 3
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AMR_2016_13
Record Dates: First submitted 2016-08-22; First posted 2016-08-29 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: HIV
MeSH Terms: interventions — elvitegravir; dolutegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- exposition to the drugs: patients treated with at least one of the following drugs: dolutegravir, elvitegravir and rilpivirine
  Interventions: Drug: prescription of at least one of the following drugs: rilpivirine, elvitegravir, dolutegravir
- patients non exposed to the drugs

INTERVENTIONS:
Drug: prescription of at least one of the following drugs: rilpivirine, elvitegravir, dolutegravir — chemical dosage ARV
  Groups: exposition to the drugs

SUMMARY:
The frequency of neurological and psychiatric complaints for participants taking rilpivirine, elvitegravir, or dolutegravir reaches on average 20-30% during clinical trials. The inclusion and exclusion criteria for enrolling people living with HIV are at times so selective and the subsequent descriptions of minor or severe adverse events (AE's) so often imprecise and ambiguous that one cannot extrapolate these particular research results to practicing medicine. These adverse events negatively affect the patient's quality of life and ultimately his or her good adherence to treatments.

This study aims at assessing the prevalence and at describing the neurological and psychiatric adverse events related to these drugs.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* age > 18
* treatment with rilpivirine, elvitegravir, or dolutegravir (for exposed patients)
* treatment with none of these drugs (for non exposed patients)
* capacity of reading French language

Exclusion Criteria:

* drugs addiction (except for amyl nitriles ("poppers") and cannabis)
* alcoholism
* co-infection with hepatitis C virus
* pregnant or breast feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients with a prescription of rilpivirine, elvitegravir, or dolutegravir (modification or initiation of an antiretroviral treatment) and non exposed HIV patients, who don't take these drugs.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
number of patients with neurologic and/or psychiatric adverse events | 6 months after modification or initiation of a treatment with one of the following drugs: dolutegravir, elvitegravir ou la rilpivirine

CONTACTS AND LOCATIONS:
Overall Officials: Antoine MOULIGNIER, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- France, Paris, France